CLINICAL TRIAL: NCT03274804
Title: A Phase I Trial of Combined PD-1 Inhibition (Pembrolizumab) and CCR5 Inhibition (Maraviroc) for the Treatment of Refractory Microsatellite Stable (MSS) Metastatic Colorectal Cancer (mCRC)
Brief Title: Combined PD-1 and CCR5 Inhibition for the Treatment of Refractory Microsatellite Stable mCRC
Acronym: PICCASSO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Responsible Party: Principal Investigator, Dirk Jäger, Prof. Dr., University Hospital Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PICCASSO
Record Dates: First submitted 2017-08-14; First posted 2017-09-07 (Actual); Results first posted 2021-04-22 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-05

CONDITIONS: Metastatic Colorectal Cancer; MSS
MeSH Terms: conditions — Colorectal Neoplasms | interventions — pembrolizumab; Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm, prospective, open-label trial (Experimental): Eligible subjects will receive pembrolizumab beginning on Day 1 of each 3-week dosing cycle (d1, qd22) together with maraviroc administered perorally on day 1 to 21 of each cycle (d1-21; qd22).
  Interventions: Biological: Pembrolizumab; Drug: Maraviroc

INTERVENTIONS:
Biological: Pembrolizumab — Eligible subjects will receive pembrolizumab beginning on Day 1 of each 3-week dosing cycle (d1, qd22)
  Other Names: Keytruda
Drug: Maraviroc — Maraviroc will be administered perorally on day 1 to 21 of each cycle (d1-21; qd22)
  Other Names: Celsentri

SUMMARY:
This is a monocentric, single arm, prospective, open-label trial of a combination treatment consisting of pembrolizumab and maraviroc in previously treated subjects who have refractory microsatellite stable (MSS) metastatic colorectal cancer (mCRC).

DETAILED DESCRIPTION:
Eligible subjects will receive pembrolizumab beginning on Day 1 of each 3-week dosing cycle (d1, qd22) together with maraviroc administered perorally on day 1 to 21 of each cycle (d1-21; qd22).

Treatment with pembrolizumab / maraviroc combination will continue until progressive disease (PD), unacceptable adverse events (AEs), intercurrent illness that prevents further administration of treatment, investigator's decision to withdraw the subject, subject withdraws consent, pregnancy of the subject, noncompliance with trial treatment or procedure requirements, administrative reasons requiring cessation of treatment, or completion of treatment per protocol.

Subjects with a treatment response or stable disease after completion of the first treatment phase of eight cycles (core treatment period) will be offered, at the discretion of the investigator, participation in a maintenance phase consisting of up to 24 additional treatment cycles of pembrolizumab monotherapy (total treatment duration up to 24 months).

Subjects who discontinue for reasons other than PD will have post-treatment follow-up for disease status until PD, initiating a non-study cancer treatment, withdrawing consent, or becoming lost to follow-up. All subjects will be followed for overall survival (OS) until death, withdrawal of consent, loss to follow-up, or the end of the study.

After the end of treatment, each subject will be followed for 30 days for AE monitoring. Serious adverse events (SAEs) and AEs of special interest (AESIs) will be collected for 90 days after the end of treatment or for 30 days after the end of treatment if the subject initiates new anticancer therapy, whichever is earlier.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic colorectal cancer. Microsatellite stability (MSS) is confirmed by PCR or immunohistochemistry.
2. Patient failed standard therapy or is intolerable towards standard therapy which must include a fluoropyrimidine, oxaliplatin, irinotecan, an antiangiogenic monoclonal antibody (e.g. bevacizumab, aflibercept, ramucirumab), an EGFR inhibitor in case of RAS/BRAF wildtype tumors and optional regorafenib or TAS 102
3. Measurable disease as per RECIST 1.1
4. Metastatic lesion accessible for repetitive biopsies and patient willing to provide tissue from newly obtained biopsies. Patients without accessible lesions might be enrolled after discussion with the principle investigator.
5. ECOG performance status 0 or 1
6. Adequate hematological, hepatic and renal function parameters:

   * Leucocytes> 3.000/μl
   * Hemoglobin >9 g/dl
   * Thrombocytes > 100.000/μl
   * Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or GFR ≥60 mL/min for subject with creatinine levels > 1.5 x institutional ULN
   * Serum total bilirubin ≤ 1.5 x upper limit of normal or direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
   * AST and ALT ≤ 2.5 x upper limit of normal (or ≤ 5 x if liver metastases are present)
   * Albumin ≥ 2.5 mg/dL
7. Adequate coagulation functions as defined by International Normalized Ratio (INR) ≤1.5, and a partial thromboplastin time (PTT) ≤ 5 seconds above the ULN (unless receiving anticoagulation therapy). Patients receiving warfarin/ phenprocoumon must be switched to low molecular weight heparin and have achieved stable coagulation profile.
8. Female and male patients' ≥ 18 years. Patients in reproductive age must be willing to use adequate contraception during the study and 4 months after the end of the study (appropriate contraception is defined as surgical sterilization (e.g., bilateral tubal ligation, vasectomy), hormonal contraception (implantable, patch, oral), and doublebarrier methods (any double combination of: IUD, male or female condom with spermicidal gel, diaphragm, sponge, cervical cap)). Abstinence (relative to heterosexual activity) can be used as the sole method of contraception if it is consistently employed as the subject's preferred and usual lifestyle and if considered acceptable by local regulatory agencies and ERCs/IRBs. Periodic abstinence (e.g., calendar, ovulation, sympto-thermal, post-ovulation methods, etc.) and withdrawal are not acceptable methods of contraception. Female patients with childbearing potential need to have a negative pregnancy test within 7 days before study start.
9. Patient able and willing to provide written informed consent and to comply with the study protocol and with the planned surgical procedures.

Exclusion Criteria:

1. Inability to understand the aims of the study and/or protocol procedures
2. Hypersensitivity towards pembrolizumab, maraviroc, or any ingredients of the formulations administered
3. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies
4. Any other concurrent antineoplastic treatment including irradiation (local radiation of single non-target lesions for palliation only allowed)
5. Active autoimmune disease requiring immunosuppressive therapy
6. Any condition requiring continuous systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 2 weeks prior to first dose of study treatment. Inhaled or topical steroids and physiological replacement doses of up to 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease.
7. Secondary malignant disease during the last 5 years (exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy).
8. Clinical relevant comorbidity also including significant psychiatric disease
9. Clinically significant active coronary heart disease, cardiomyopathy or congestive heart failure, NYHA III-IV
10. Cardiocirculatory insufficiency with hypotension (systolic blood pressure <100 mmHg)
11. Cirrhosis of the liver (Child > Grade A), pronounced alcohol abuse with anticipated detoxification, severe pulmonary infection with considerable reduction of pulmonary function
12. Prior allogeneic bone marrow transplantation
13. Prior treatment with anti-PD-1, anti-PD-L1, or anti-PD-L2 therapeutic antibody
14. Administration of a live, attenuated vaccine within four weeks prior to start of maintenance treatment or anticipation that such a live attenuated vaccine will be required during the remainder of the study Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
15. Chronic intake of drugs that lead to known interference with Maraviroc metabolism through strong Cytochrome P450 3A4 (CYP3A4) interaction: e.g. Rifampicin, Rifabutin, Clarithromycin, Telithromycin, Ketoconazole, Itraconazole, Fluconazole, Hypericum perforatum (St. John's Worth /Johanniskraut) or any strong CYP3A4 inducing or inhibiting drug (See Section 5.5.2)
16. Positive test for human immunodeficiency virus (HIV) or HIV infection
17. Active hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test) or hepatitis C. Note: Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen antibody test) are eligible.
18. Active or latent tuberculosis
19. Clinically active brain metastases, defined as untreated symptomatic, or requiring therapy with steroids or anticonvulsants to control associated symptoms.

    Subjects with treated brain metastases that are no longer symptomatic and require no treatment with steroids may be included in the study if they have recovered from the acute toxic effect of radiotherapy and have no evidence of disease progression on imaging studies (MRI/CT scan).
20. On-treatment participation in another clinical study in the period 30 days prior to start of study treatment and during the study
21. Patients in a closed institution according to an authority or court decision (AMG § 40, Abs. 1 No. 4)
22. Pregnancy or lactation
23. Known history of, or any evidence of active, non-infectious pneumonitis or interstitial lung disease.
24. Active infection requiring systemic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Jäger, Prof., Principal Investigator — NCT, Med Oncology, University Hospital Heidelberg
Locations (1):
- National Center for Tumor Diseases, University Hospital Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haag GM, Springfeld C, Grun B, Apostolidis L, Zschabitz S, Dietrich M, Berger AK, Weber TF, Zoernig I, Schaaf M, Waberer L, Muller DW, Al-Batran SE, Halama N, Jaeger D. Pembrolizumab and maraviroc in refractory mismatch repair proficient/microsatellite-stable metastatic colorectal cancer - The PICCASSO phase I trial. Eur J Cancer. 2022 May;167:112-122. doi: 10.1016/j.ejca.2022.03.017. Epub 2022 Apr 12. PMID 35427833

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm, Prospective, Open-label Trial
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The required parameters as defined in the inclusion and exclusion criteria are met by all patients.
Groups:
- Study Treatment Arm: All enrolled subjects received pembrolizumab 200 mg IV on day one every three weeks (d1, qd22; Q3W) plus maraviroc 2 x 300 mg p.o. daily as combination therapy in an unblinded fashion.
Arm/Group | Study Treatment Arm
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 9
Age, Continuous [Median (Standard Deviation); unit: years] | 61 (8.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 20

OUTCOME MEASURES:

1. Primary Outcome: Feasibility Rate of a Combined Therapy
Description: Defined as the rate of patients receiving the protocol treatment according to the planned schedule without occurrence of at least one of the following events:
  Study treatment-related Grade ≥ 3 immune-related abnormalities; Study treatment-related Grade ≥ 4 AEs of any aetiology; Any toxic event leading to the premature withdrawal of protocol treatment
Time Frame: After core treatment period of 8 cycles (each cycle is 21 days)
Measure: Count of Participants; unit: Participants
Groups:
- Single Arm, Prospective, Open-label Trial: All enrolled subjects received pembrolizumab 200 mg IV on day one every three weeks (d1, qd22; Q3W) plus maraviroc 2 x 300 mg p.o. daily as combination therapy in an unblinded fashion.
Arm/Group | Single Arm, Prospective, Open-label Trial
Number analyzed (Participants) | 19
Participants | 18

2. Secondary Outcome: Safety and Toxicity of a Combined Therapy Based on Subjects Who Experienced Toxicities
Description: The primary safety analysis will be based on subjects who experienced toxicities as defined by the current National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE, v4.0; Section 11.2). The attribution to drug, time-of-onset, duration of the event, its resolution, and any concomitant medications administered will be recorded.
Time Frame: After core treatment period of 8 cycles (each cycle is 21 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Study Treatment Arm
Number analyzed (Participants) | 20
Participants | 20

3. Secondary Outcome: Efficacy Endpoint: Disease Control Rate
Description: Determine DCR defined as percentage of patients displaying CR/PR or SD as best response according to the RECIST criteria version 1.1.
Time Frame: through study completion (20 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Study Treatment Arm
Number analyzed (Participants) | 19
Participants | 1

4. Secondary Outcome: Efficacy Endpoint: Objective Response Rate
Description: ORR and immune related (ir) ORR (irORR) will be analyzed.
Time Frame: through study completion (20 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm, Prospective, Open-label Trial
Number analyzed (Participants) | 19
Participants | 1

5. Secondary Outcome: Efficacy Endpoint: Progression-free Survival
Description: Individual PFS will be analyzed.
Time Frame: through study completion (20 months)
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Study Treatment Arm
Number analyzed (Participants) | 19
weeks | 9 [7.00 to 10.00]

6. Secondary Outcome: Overall Survival
Description: Individual OS will be analyzed.
Time Frame: through study completion (20 months)
Measure: Median (95% Confidence Interval); unit: Time until event, month
Arm/Group | Study Treatment Arm
Number analyzed (Participants) | 19
Time until event, month | 9 [6.00 to 20.00]

ADVERSE EVENTS:
Time Frame: From the time of treatment allocation through 30 days following discontinuation of treatment, up to 20 months, all adverse events must be reported by the investigator.
Groups:
- Study Treatment Arm: The primary safety analysis will be based on subjects who experienced toxicities as defined by the current National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE, v4.0; Section 11.2). The attribution to drug, time-of-onset, duration of the event, its resolution, and any concomitant medications administered will be recorded.
Arm/Group | Study Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 4/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Treatment Arm (N=20)
Infections and infestations - Other (Infections and infestations) | 1 (1) — unknown origin
Catheter related infection (Infections and infestations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study Treatment Arm (N=20)
Abdominal pain (Gastrointestinal disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Anal hemorrhage (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1
Blood bilirubin increased (Investigations) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Bronchial infection (Infections and infestations) | 1
Catheter related infection (Infections and infestations) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Chills (General disorders) | 1
Conjunctivitis (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Creatinine increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1
Edema limbs (General disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 1
Fatigue (General disorders) | 1
Fever (General disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Flushing (Vascular disorders) | 1
Gallbladder obstruction (Hepatobiliary disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 1
Headache (Nervous system disorders) | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1
Hot flashes (Vascular disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Insomnia (Psychiatric disorders) | 1
Investigations - Other, specify (Investigations) | 1
Keratitis (Eye disorders) | 1
Localized edema (General disorders) | 1
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Nail infection (Infections and infestations) | 1
Nausea (Gastrointestinal disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Rash pustular (Infections and infestations) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1
Salivary gland infection (Infections and infestations) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Stomach pain (Gastrointestinal disorders) | 1
Tooth infection (Infections and infestations) | 1
Tremor (Nervous system disorders) | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Urinary frequency (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 1
Weight gain (Investigations) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT03274804/Prot_SAP_000.pdf